CLINICAL TRIAL: NCT05141669
Title: Impact of Fingolimod Adherence on Outcomes
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CFTY720DUS45
Record Dates: First submitted 2021-11-19; First posted 2021-12-02 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fingolimod: Participants who initiated fingolimod to treat multiple sclerosis (MS)
  Interventions: Drug: Fingolimod
- Non-fingolimod Disease Modifying Treatment (DMT): All patients with ≥ 1 medical or pharmacy claim for a DMT other than fingolimod. Among patients included in the study that those with ≥ 1 pharmacy or medical claim for any MS DMT during pre-index would be excluded.

INTERVENTIONS:
Drug: Fingolimod — Participants who initiated fingolimod to treat multiple sclerosis (MS)
  Groups: Fingolimod

SUMMARY:
This study was a retrospective observational claims data study of commercial and Medicare Advantage with Part D (MAPD) patients initiating fingolimod.

DETAILED DESCRIPTION:
The study sample comprised commercial and MAPD enrollees who initiated fingolimod treatment during the identification period of 01 January 2012 through 10 May 2018. The date of the first fingolimod pharmacy claim during the identification period was the index date.

All patients were continuously enrolled in the health plan for 24 months. The 6-month pre-index period, ending the day before the index date, was used to assess patients' clinical characteristics (e.g., comorbid conditions and MS symptoms). The 18-month post-index period started on the index date. The first 6 months of the post-index period (initiation period) were used to assess MS symptoms and adherence. Months 7 - 18 of the post-index period (post-initiation period) were used to measure adherence and outcomes. The 24-month observation period for each patient comprised the 6-month pre-index and 18-month post-index periods.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old during year of index date with valid gender and geographic information
* Continuous enrollment (CE) in the health plan with medical and pharmacy benefits for ≥6 months (180ii days) before the index date (pre-index period)
* CE with medical and pharmacy benefits for ≥18 months (540 days) beginning on the index date (post-index period)

  * All patients had uniform 6-month pre-index and 18-month post-index periods
* ≥1 medical claim with an MS diagnosis codei in any position during the pre-or post-index periods
* ≥1 claim for fingolimod after the index date (i.e., from index date +1 to 539 days post-index)

  * By requiring ≥1 medical claim with an MS diagnosis code and ≥2 claims with an NDC for fingolimod, the inclusion criteria essentially incorporated the preferred/overall best performing MS case-finding definition validated by Culpepper et al. The criteria for that definition required at least 3 separate encounters from any of the following: MS-related ambulatory visits, MS-related inpatient stays, and DMT claims during a 12-month period. Slightly higher accuracy was found when a 24-month period was used.

Exclusion Criteria:

•≥1 pharmacy or medical claim for any MS DMT during the pre-index period

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study comprised of commercial and Medicare Advantage with Part D (MAPD) enrollees who initiated fingolimod treatment during the identification period of 01 January 2012 through 10 May 2018.
Sampling Method: Non-Probability Sample
Enrollment: 694 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
Number of Multiple Sclerosis (MS) relapses | Month 7 to Month 18 (12 months) of the post-index period. The date of the first fingolimod claim was the index date (01 January 2012 through 10 May 2018)
  Number of Multiple Sclerosis (MS) relapses were reported to estimate the effect of fingolimod adherence on the odds of MS relapse in a 12-month period

SECONDARY OUTCOMES:
Number of Multiple Sclerosis-related inpatient admission | Month 7 to Month 18 (12 months) of the post-index period. The date of the first fingolimod claim was the index date (01 January 2012 through 10 May 2018)
  Number of any Multiple Sclerosis-related inpatient admission were reported to estimate the effect of fingolimod adherence during a 12 month period for Disease Modifying Treatment (DMT) treatment-naïve adult MS patients in the commercial and MAPD populations.
Number of Multiple Sclerosis-related Emergency Room (ER) visits | Month 7 to Month 18 (12 months) of the post-index period. The date of the first fingolimod claim was the index date (01 January 2012 through 10 May 2018)
  Number of Multiple Sclerosis-related ER visits were reported to estimate the effect of fingolimod adherence during a 12 month period for Disease Modifying Treatment (DMT) treatment-naïve adult MS patients in the commercial and MAPD populations.
All-cause total (medical plus pharmacy) health care costs | Month 7 to Month 18 (12 months) of the post-index period. The date of the first fingolimod claim was the index date (01 January 2012 through 10 May 2018)
  All-cause total (i.e., pharmacy + medical costs) were computed as the combined health plan and patient paid amounts for all claims, regardless of diagnoses recorded. Medical costs comprised sub-categories of ambulatory costs (physician office and hospital outpatient), emergency services costs, inpatient costs, and other medical costs.
All-cause medical health care costs | Month 7 to Month 18 (12 months) of the post-index period. The date of the first fingolimod claim was the index date (01 January 2012 through 10 May 2018)
  Medical health care costs were reported to estimate the effect of fingolimod adherence during a 12 month period for Disease Modifying Treatment (DMT) treatment-naïve adult MS patients in the commercial and MAPD populations.
All-cause total (medical plus pharmacy) health care costs excluding fingolimod | Month 7 to Month 18 (12 months) of the post-index period. The date of the first fingolimod claim was the index date (01 January 2012 through 10 May 2018)
  Total (medical plus pharmacy) health care costs excluding fingolimod were reported to estimate the effect of fingolimod adherence during a 12 month period for Disease Modifying Treatment (DMT) treatment-naïve adult MS patients in the commercial and MAPD populations.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigational Site, East Hanover, New Jersey, United States

REFERENCES:
- See also: Results for CFTY720DUS45 from the Novartis Clinical Trials Website — http://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17883